CLINICAL TRIAL: NCT00058279
Title: MDX-CTLA4 Combined With IL-2 for Patients With Metastatic Melanoma
Brief Title: Monoclonal Antibody Therapy and Interleukin-2 in Treating Patients With Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000287211; NCI-03-C-0109; NCT00055211 (obsolete NCT alias)
Record Dates: First submitted 2003-04-07; First posted 2003-04-09 (Estimated); Last update posted 2013-06-20 (Estimated); Status verified 2006-08

CONDITIONS: Intraocular Melanoma; Melanoma (Skin)
Keywords: stage IV melanoma; extraocular extension melanoma; recurrent melanoma; iris melanoma; ciliary body and choroid melanoma, medium/large size; ciliary body and choroid melanoma, small size; recurrent intraocular melanoma
MeSH Terms: conditions — Uveal Melanoma; Melanoma | interventions — aldesleukin; Ipilimumab

INTERVENTIONS:
Biological: aldesleukin
Biological: ipilimumab

SUMMARY:
RATIONALE: Biological therapies, such as MDX-010, work in different ways to stimulate the immune system and stop tumor cells from growing. Interleukin-2 may stimulate a person's white blood cells to kill tumor cells. Combining monoclonal antibody therapy with interleukin-2 may kill more tumor cells.

PURPOSE: Phase I/II trial to study the effectiveness of combining monoclonal antibody therapy with interleukin-2 in treating patients who have metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose (MTD) of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-CTLA4) in combination with high-dose interleukin-2 (IL-2) in patients with metastatic melanoma. (Phase I is closed to accrual as of 4/13/2004).
* Determine the activity of MDX-CTLA4 administered at the MTD with high-dose IL-2 in these patients.
* Determine whether the administration of IL-2 alters the pharmacokinetics of MDX-CTLA4 in these patients.
* Determine the safety and adverse event profile of this regimen in these patients.

OUTLINE: This is an open-label, dose-escalation study of anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-CTLA4).

* Phase I: Patients receive MDX-CTLA4 IV on days 0, 21, and 42. Patients also receive high-dose interleukin-2 (IL-2) IV over 15 minutes every 8 hours for up to 15 doses beginning on days 22 and 43. Treatment repeats every 63 days for up to 3 courses in the absence of disease progression or unacceptable toxicity. Patients with an ongoing partial response and no greater than grade 1 toxicity may receive additional courses of therapy. Patients who require discontinuation of MDX-CTLA4 due to toxicity may continue receiving IL-2 at the discretion of the investigator.

Cohorts of 3-6 patients receive escalating doses of MDX-CTLA4 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. (Phase I is closed to accrual as of 4/13/2004).

* Phase II: Patients receive treatment as in phase I at the MTD of MDX-CTLA4. Patients who achieve a partial or complete response and later develop recurrent or progressive disease may be retreated at the same dose.

Patients are followed at 3 weeks, every 3 months for 1 year, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 3-51 patients (3-18 for phase I and 19-33 for phase II) will be accrued for this study within 1 year. (Phase I is closed to accrual as of 4/13/2004).

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage IV melanoma

  * Mucosal or ocular melanoma also eligible
* Clinically evaluable disease

  * At least 1 site of measurable disease

PATIENT CHARACTERISTICS:

Age

* 16 and over

Performance status

* ECOG 0-1

Life expectancy

* At least 3 months

Hematopoietic

* WBC at least 2,500/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10 g/dL
* Hematocrit at least 30%

Hepatic

* Bilirubin no greater than upper limit of normal (ULN)* (less than 3.0 mg/dL in patients with Gilbert's syndrome)
* AST no greater than 3 times ULN*
* Hepatitis B surface antigen negative
* Hepatitis C antibody nonreactive
* No evidence or history of significant hepatic disease that would preclude safe administration of high-dose IL-2 NOTE: *Unless attributable to disease

Renal

* Creatinine no greater than 2.0 mg/dL
* No evidence or history of significant renal disease that would preclude safe administration of high-dose IL-2

Cardiovascular

* No evidence or history of significant cardiac disease that would preclude safe administration of high-dose IL-2
* Thallium stress test normal (for patients over 50 years of age or with a history of cardiovascular disease)

Pulmonary

* No evidence or history of significant pulmonary disease that would preclude safe administration of high-dose IL-2

Immunologic

* HIV negative
* No autoimmune disease (including uveitis and autoimmune inflammatory eye disease)
* No active infection

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except adequately treated basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the cervix
* No evidence or history of significant gastrointestinal disease that would preclude safe administration of high-dose IL-2
* No evidence or history of psychiatric disease that would preclude safe administration of high-dose IL-2
* No other underlying medical condition that would make the administration of the study drug hazardous or obscure the interpretation of adverse events
* No other concurrent medical condition that would preclude study entry

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 3 weeks since prior immunotherapy for melanoma and recovered
* No prior anti-cytotoxic T-lymphocyte-associated antigen-4 monoclonal antibody (MDX-CTLA4)
* No prior high-dose (at least 600,000 IU/kg every 8 hours) interleukin-2 (IL-2)

Chemotherapy

* At least 3 weeks since prior chemotherapy for melanoma and recovered
* No concurrent chemotherapy

Endocrine therapy

* At least 3 weeks since prior hormonal therapy for melanoma and recovered
* At least 4 weeks since prior corticosteroids
* No concurrent systemic or topical corticosteroids

Radiotherapy

* At least 3 weeks since prior radiotherapy for melanoma and recovered

Surgery

* Not specified

Other

* No concurrent immunosuppressive agents (e.g., cyclosporine or its analog)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2003-02; Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steven A. Rosenberg, MD, PhD, Study Chair — NCI - Surgery Branch
Locations (1):
- Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland, United States

REFERENCES:
- [Result] Maker AV, Phan GQ, Attia P, Yang JC, Sherry RM, Topalian SL, Kammula US, Royal RE, Haworth LR, Levy C, Kleiner D, Mavroukakis SA, Yellin M, Rosenberg SA. Tumor regression and autoimmunity in patients treated with cytotoxic T lymphocyte-associated antigen 4 blockade and interleukin 2: a phase I/II study. Ann Surg Oncol. 2005 Dec;12(12):1005-16. doi: 10.1245/ASO.2005.03.536. Epub 2005 Oct 21. PMID 16283570
- [Derived] Schadendorf D, Hodi FS, Robert C, Weber JS, Margolin K, Hamid O, Patt D, Chen TT, Berman DM, Wolchok JD. Pooled Analysis of Long-Term Survival Data From Phase II and Phase III Trials of Ipilimumab in Unresectable or Metastatic Melanoma. J Clin Oncol. 2015 Jun 10;33(17):1889-94. doi: 10.1200/JCO.2014.56.2736. Epub 2015 Feb 9. PMID 25667295